CLINICAL TRIAL: NCT04881669
Title: The Effect of the Wall Thickness of Obturator Bulbs on Masticatory Function in Patients With Maxillectomy
Brief Title: The Effect of Obturator Thickness on the Function
Acronym: obturator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dr. Merve Benli, Assistant Professor, Istanbul University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1297
Record Dates: First submitted 2021-05-03; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Maxilla--Cancer
Keywords: obturator, bulb

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low group (Experimental): low thickness group
  Interventions: Device: obturator
- moderate group (Experimental): moderate thickness group
  Interventions: Device: obturator
- high group (Experimental): high thickness group
  Interventions: Device: obturator

INTERVENTIONS:
Device: obturator — variable bulbs
  Other Names: bulb

SUMMARY:
the effect of obturator bulb thickness on masticatory function has been verified.

ELIGIBILITY:
Inclusion Criteria:

* having maxillectomy operation

Exclusion Criteria:

* having radiation therapy before the study

Ages: 16 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
the effect of bulb thickness | 3 weeks
  measuring the efficacy of masticatory function with chewing test
the effect of weight reduction | 3 weeks
  measuring the weight differences of prostheses

CONTACTS AND LOCATIONS:
Overall Officials: merve benli, phd, Study Director — Istanbul University
Locations (1):
- Istanbul university,Faculty of Dentistry, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol